CLINICAL TRIAL: NCT01283412
Title: Intraoperative Application of Dexmedetomidine on the Incidence of Postoperative Delirium and Quality of Recovery in Geriatric Patients Undergoing Major Surgery
Brief Title: Dexmedetomidine on Postoperative Delirium and Quality of Recovery in Geriatric Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Associate Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIHMZK02004
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Delirium, Postoperative
Keywords: Delirium; Dexmedetomidine; Adult Patients; Elective Major Surgery; General Anesthesia
MeSH Terms: conditions — Emergence Delirium; Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm P (Active Comparator): Placebo infusion
  Interventions: Drug: Placebo
- Arm D (Experimental): Dexmedetomidine infusion
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Placebo — Placebo (saline) iv. during the operation and stoped 30min before end of the surgery
  Arms: Arm P
Drug: Dexmedetomidine — Dexmedetomidine 0.1~0.2ug/kg/h iv. during the operation, and stoped 30min before end of surgery
  Arms: Arm D

SUMMARY:
Postoperative agitation (hyperactive delirium) is common following major surgery(incidence was about 20% in our pilot study). Dexmedetomidine was related to a reduced delirium rate when comparing with midazolam in many clinical settings. It is not clear if dexmedetomidine is useful on reducing postoperative delirium. The hypothesis of present study: intraoperative application of dexmedetomidine (0.2ug/kg/h) is is effective (50% reduce) than placebo for reducing of early postoperative delirium and increase postoperative quality of recovery within 24 postoperative hours.

DETAILED DESCRIPTION:
After approval from the Institute's Ethics Committee, this study was conducted at Tongji Hospital, a general university teaching hospital with 2500 beds in Wuhan, China.The study consisted of adult patients, American Society of Anaesthesiologists Physical Status (ASA-PS) I-III, undergoing selective major surgery under general anesthesia. All the patients were randomly assigned to receive dexmedetomidine or placebo during the operation. The primary outcome measure was postoperative delirium assessed by Nursing Delirium Screening Scale (Nu-DESC) every 8 hours within 24 postoperative hours. The secondary outcome was length of postanesthesia care unit (PACU) stay,postoperative hospital length of stay, hemodynamic parameters, the incidence of postoperative nausea and vomiting, and quality of recovery determined by quality of recovery (QOR40; maximum score 200)and Post-operative Quality Recovery Scale (PQRS) in the first 24 h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class I-III
* Aged 60 years or above
* Elective major surgery under general anesthesia

Exclusion Criteria:

* ASA-PS>=IV
* Aged under 60 yr old
* Body mass index (BMI) >30
* Neurologic disease
* Cardiac surgery and neurologic surgery
* Anticonvulsant drugs
* Chronic analgesics intake
* Participating in the investigation of another study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | every 8 hours within 24 postoperative hours
  Postoperative delirium was determined by Nu-DESC every 8 hours within 24 postoperative hours

SECONDARY OUTCOMES:
Length of PACU stay | during PACU stay
  Length of PACU stay (min)
hemodynamic parameters | every 5min during operation and every 15min during PACU stay
  Heart frequency, systolic blood pressure, diastolic blood pressure
incidence of postoperative nausea and vomiting | 24 postoperative hours
  incidence of postoperative nausea and vomiting
quality of recovery determined by QOR40 and Postoperative Quality Recovery Scale (PQRS) | 24 postoperative hours
  quality of recovery determined by QOR40 and Postoperative Quality Recovery Scale (PQRS)
Postoperative delirium | 1st, 2nd, 3rd postoperative days
  Postoperative delirium was determined by Nu-DESC every 8 hours within 24 postoperative hours
Postoperative Stroke | 1st, 2nd, 3rd, 7th postoperative days
  Postoperative Stroke will be determined by National Institute of Health stroke scale (NIHSS score).

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, M.D., Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology; Chuanhan Zhang, MD., Study Director — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China